CLINICAL TRIAL: NCT05289895
Title: Clinical Study on Prognostic Biomarkers of Pancreatic Cancer Based on Proteomic Technique
Brief Title: Prognostic Biomarkers of Pancreatic Cancer Based on Proteomic Techniques
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: JJDB-SR-2021-04
Record Dates: First submitted 2022-03-06; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Proteomics; Pancreatic Cancer; Prognostic Biomarkers
Keywords: proteomics; Pancreatic Cancer; Prognostic Biomarkers
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Sequence I (Retrospective study: proteomic analysis of pathological specimens and information collection of previous patients with pancreatic cancer)
  Interventions: Other: No intervention
- 2: Sequence 2 (Non-interventional prospective study, sample and information collection in patients with pancreatic cancer)
  Interventions: Other: No intervention
- 3: Sequence 3 (Non-intervention study, healthy subjects sample and information collection)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This study was an observational trial without any intervention

SUMMARY:
Sequence I (Retrospective study: proteomic analysis of pathological specimens and information collection of previous patients with pancreatic cancer) Sequence 2 (Non-interventional prospective study, sample and information collection in patients with pancreatic cancer) Sequence 3 (Non-intervention study, healthy subjects sample and information collection)

DETAILED DESCRIPTION:
Sequence 1 was a retrospective study, which collected pathological tissue samples (continuous cut white slices, 10 slices per case, 2 of which were HE stained slices) and clinical data (including clinical diagnostic information, laboratory examination results, imaging findings, and prognosis information) from 100 patients with pancreatic cancer. Proteomic analysis was performed on the samples. Sequence 2 was a non-intervention prospective study, which would collect pathological tissue samples (continuous cut white slices, 10 slices per case, 2 of which were hematoxylin-eosin staining (HE) stained slices) , blood (4ml ) and urine (5mL) samples from 100 subjects with pancreatic cancer before medication. The pathological samples and clinical information of the subjects were collected for proteomic analysis. Sequence 3 was a non-intervention study, which would collect blood (4ml ) and urine (5mL) samples from 20 healthy subjects (as control samples for proteomic analysis)

ELIGIBILITY:
Inclusion Criteria:

Sequence 1 (pathological specimens and information collection of pancreatic cancer patients):

1. Chinese patients, regardless of age and gender;
2. patients with pancreatic cancer confirmed by pathology;
3. Patients without a second primary tumor;
4. The clinical diagnostic information to be collected within three months before sampling is relatively complete.

Sequence 2 (samples and information collection of patients with pancreatic cancer):

1. Chinese patients, regardless of age and gender;
2. Subjects must obtain informed consent and sign informed consent, indicating that they understand the purpose and procedure of this study and are willing to participate in the study;
3. Patients with pancreatic malignancy diagnosed by pathology;
4. Patients without a second primary tumor.

Sequence 3 (healthy subject samples and information collection)

1. Chinese healthy male or female, aged 18-45;
2. Subjects must obtain informed consent and sign informed consent, indicating that they understand the purpose and procedure of this study and are willing to participate in the study;
3. Physical examination, vital signs, laboratory examination (blood routine, blood biochemistry and urine routine), 12 lead ECG and other normal or abnormal persons without clinical significance

Exclusion Criteria:

Sequence 1 :

1. The quality of pathological specimens of patients can not meet the requirements of proteomics;
2. The researchers believe that patients who are not suitable for proteomic analysis.

Sequence 2:

1. patients with other malignant tumors (non pancreatic cancer metastasis).
2. hepatitis B surface antigen positive, hepatitis C antibody positive, HIV antibody positive or syphilis antibody positive;
3. Pregnant or lactating women;
4. The researcher believes that it is not suitable to participate in this experiment.

Sequence 3:

1. Abnormalities of clinical significance judged by clinicians, including physical examination, vital signs examination, ECG or clinical laboratory examination results;
2. hepatitis B surface antigen positive, hepatitis C antibody positive, HIV antibody positive or syphilis antibody positive;
3. Those who have participated in other clinical trials of drugs and accepted clinical trials of drugs or devices for trial within the first three months;
4. Those vaccinated with active or attenuated vaccine within 1 month before screening or during the planned trial;
5. Pregnant or lactating women;
6. Those who have taken any drugs within the first 14 days;
7. The researcher believes that it is not suitable to participate in this experiment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healty Chinese volunteers and Pancreatic cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Proteomic analysis of tumor tissue samples | 2 years
  Proteomic analysis of tumor tissue samples from patients with pancreatic cancer
Proteomic analysis of blood and urine | 1 year
  Proteomic analysis of blood and urine in healthy volunteers and patients with pancreatic cancer

IPD SHARING:
Plan to Share IPD: No
This study is confidential. All the technical achievements and outcomes of this trial are owned by the Affiliated Hospital of Qingdao University and two two cooperative research organization.